CLINICAL TRIAL: NCT02806375
Title: Graft-versus-host Disease Prophylaxis With Post-transplantation Cyclophosphamide and Ruxolitinib in Patients With Myelofibrosis
Brief Title: PTCy and Ruxolitinib GVHD Prophylaxis in Myelofibrosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: St. Petersburg State Pavlov Medical University (Other)
Responsible Party: Principal Investigator, Ivan S Moiseev, Vice-director for science of R.M. Gorbacheva Memorial Institute of Hematology, Oncology and Transplantation, St. Petersburg State Pavlov Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04/16-n
Record Dates: First submitted 2016-06-08; First posted 2016-06-20 (Estimated); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Primary Myelofibrosis; Myeloproliferative Disorders
Keywords: Myelofibrosis; Ruxolitinib; Cyclophosphamide; Immunosuppressive Agents; Immune System Diseases; Busulfan; Fludarabine; Antineoplastic Agents, Alkylating; Myeloablative Agonists; Hematopoietic Stem Cell Transplantation; Allogeneic
MeSH Terms: conditions — Primary Myelofibrosis; Myeloproliferative Disorders; Immune System Diseases | interventions — Busulfan; fludarabine phosphate; Cyclophosphamide; ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- PTCy and ruxolitinib (Experimental)
  Interventions: Procedure: Allogeneic hematopoietic stem cell transplantation; Drug: Busulfan; Drug: Fludarabine monophosphate; Drug: Cyclophosphamide; Drug: Ruxolitinib

INTERVENTIONS:
Procedure: Allogeneic hematopoietic stem cell transplantation — Day 0: Infusion of unmanipulated graft
  Other Names: HSCT
Drug: Busulfan — Days -5 through -3: Busulfan 1 mg/kg po qid №10
Drug: Fludarabine monophosphate — Days -7 through -2: 30 mg/m2/day iv qd x 6 days
Drug: Cyclophosphamide — Day +3 and +4: 50 mg/kg/day iv qd
  Other Names: Cytoxan
Drug: Ruxolitinib — Days -8 through -2 15 mg tid
Drug: Ruxolitinib — Days +5 through +100: 7.5 mg bid

SUMMARY:
A number of groups have demonstrated very low incidence of acute and chronic graft-versus-host disease (GVHD) with post-transplantation cyclophosphamide (PTCy) in haploidentical and unrelated allogeneic stem cell transplantation (SCT). Still the relapse of the underlining malignancy is a problem after this prophylaxis. Ruxolitinib is currently one of the most promising drugs in the treatment of steroid-refractory GVHD. On the other hand, its primary indication is myelofibrosis, and it was demonstrated that ruxolitinib before allogeneic SCT might improve the outcome. This pilot trial evaluates whether the combination of PTCy and ruxolitinib facilitates adequate GVHD control, and decreases the risk of graft failure and disease progression in myelofibrosis patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have an indication for allogeneic hematopoietic stem cell transplantation
* Diagnosis:

Primary myelofibrosis Secondary myelofibrosis

* Signed informed consent
* Matched related, 8-10/10 HLA-matched unrelated or haploidentical donor available. The HLA typing is performed by the following genetic loci: HLA-A, HLA-B, HLA-Cw, HLA-DRB1, and HLA-DQB1.
* No second tumors
* No severe concurrent illness

Exclusion Criteria:

* Moderate or severe cardiac dysfunction, left ventricular ejection fraction <50%
* Moderate or severe decrease in pulmonary function, FEV1 <70% or DLCO<70% of predicted
* Respiratory distress >grade I
* Severe organ dysfunction: AST or ALT >5 upper normal limits, bilirubin >1.5 upper normal limits, creatinine >2 upper normal limits
* Creatinine clearance < 60 mL/min
* Uncontrolled bacterial or fungal infection at the time of enrollment
* Requirement for vasopressor support at the time of enrollment
* Karnofsky index <30%
* Pregnancy
* Somatic or psychiatric disorder making the patient unable to sign informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
Incidence of acute graft-versus-host disease, grades II-IV | 180 days
Incidence of chronic GVHD, moderate and severe (NIH criteria) | 365 days

SECONDARY OUTCOMES:
Incidence of primary or secondary graft failure | 60 days
Non-relapse mortality analysis | 365 days
  Non-relapse mortality is defined as any death in absence of relapse or progressive disease. Summarized using Kaplan-Meier and cumulative incidence estimates.
Overall survival analysis | 365 days
  Summarized using Kaplan-Meier and cumulative incidence estimates.
Event-free survival analysis | 365 days
  Event is defined as relapse or death in the specified time frame. Summarized using Kaplan-Meier and cumulative incidence estimates.
Relapse rate analysis | 365 days
  Summarized using Kaplan-Meier and cumulative incidence estimates.
Number of participants with treatment-related adverse events as assessed by CTCAE v4.03 | 100 days
  Toxicity parameters based on NCI CTCAE 4.03 grades: hepatotoxicity (liver function tests), nephrotoxicity (creatinine), neurotoxicity (attending physician assessment), mucositis (attending physician assessment), hemorrhagic cystitis (attending physician assessment), cardiotoxicity (ECG, echocardiography). Additional toxicity parameters: incidence and severity of veno-occlusive disease, incidence of transplant-associated microangiopathy
Infectious complications, including analysis of severe bacterial, fungal and viral infections incidence | 100 days

CONTACTS AND LOCATIONS:
Overall Officials: Boris V. Afanasyev, Professor, Study Director — St. Petersburg State Pavlov Medical University
Locations (1):
- First Pavlov State Medical University of St. Petersburg, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: Undecided
Consultations with lawyers are ongoing about how IPD initiative fits the local law "About personal data 152-fz".

REFERENCES:
- [Derived] Morozova EV, Barabanshikova MV, Moiseev IS, Shakirova AI, Barhatov IM, Ushal IE, Rodionov GG, Moiseev SI, Surkova EA, Lapin SV, Vlasova JJ, Rudakova TA, Darskaya EI, Baykov VV, Alyanski AL, Bondarenko SN, Afanasyev BV. A Prospective Pilot Study of Graft-versus-Host Disease Prophylaxis with Post-Transplantation Cyclophosphamide and Ruxolitinib in Patients with Myelofibrosis. Acta Haematol. 2021;144(2):158-165. doi: 10.1159/000506758. Epub 2020 Apr 23. PMID 32325461